CLINICAL TRIAL: NCT05621551
Title: Effects of Perioperative Dapagliflozin on Type 2 Diabetic Patients Undergoing Cardiac Surgery
Brief Title: Dapagliflozin Therapy In Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-1437
Record Dates: First submitted 2022-11-04; First posted 2022-11-18 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2; Cardiac Surgery
Keywords: SGLT2 inhibitors; Cardiac Surgery; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin 10 mg
  Interventions: Drug: Dapagliflozin
- Standard of care (No Intervention): Standard care treatment of diabetes patients during perioperative cardiac surgery in our center

INTERVENTIONS:
Drug: Dapagliflozin — The patients is required to receive dapagliflozin(10mg, q.d.) at least for 3 days until 24 hours before the surgery. Then dapagliflozin will be discontinued and recovered as soon as the patient is able to take oral diet postoperatively. Dapagliflozin wil be ceased five days after surgery.
  Arms: Dapagliflozin

SUMMARY:
This randomized controlled trial is to assess the effects of perioperative dapagliflozin on type 2 diabetic patients undergoing cardiac surgery

DETAILED DESCRIPTION:
Sodium-Glucose Cotransporter 2 Inhibitor(SGLT2i) including dapagliflozin are widely used in the clinical treatment of type 2 diabetes mellitus(T2DM). In recent studies, SGLT2i were found to not only reduce blood glucose but also protect the heart and kidney, which can significantly reduce cardiovascular events, delay the progression of renal failure, greatly improve the quality of life of patients. Patients with T2DM have poorer cardiac surgery outcomes compared with non-diabetics. Based on the promising pharmacological profile of dapagliflozin, we hypothesize that perioperative dapagliflozin therapy would improve postoperative outcomes among patients undergoing cardiac surgery with T2DM. This randomized controlled trial is to assess the effects of perioperative dapagliflozin on type 2 diabetic patients undergoing cardiac surgery

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at screening
2. Scheduled for cardiac surgery (on-pump coronary artery bypass grafting, aortic valve replacement, or a combination of both)
3. Diagnosis of Type 2 Diabetes
4. Provision of signed informed consent prior to any study specific procedures

Exclusion Criteria:

1. Emergency surgery and non-primary surgery
2. Moderate and severe dehydration; systolic pressure≤90mmHg; unstable haemodynamics
3. History of diabetic ketoacidosis; type 1 diabetes mellitus
4. Receiving therapy with an SGLT2 inhibitor within 4 weeks prior to enrolment
5. Known allergy or hypersensitivity to dapagliflozin or other SGLT-2 inhibitors
6. Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2 or requiring dialysis; unstable or rapidly progressing renal disease at the time of randomisation
7. Serious hepatic disease
8. Women who are pregnant, nursing, or who plan to become pregnant while in the trial
9. Currently enrolled in another investigational drug study, or less than 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Hs-Troponin-I | within 2 days after surgery
  high sensitive cardiac troponin-I

SECONDARY OUTCOMES:
Renal function | within 5 days after surgery
  Acute kidney injury determined by creatinine changes and the need for renal replacement therapy, along with creatinine changes and the need for renal replacement therapy themselves.
NT-proBNP | within 5 days after surgery
  N-terminal prohormone of brain natriuretic peptide
Postoperative atrial fibrillation | within 5 days after surgery
  In this study, postoperative AF was defined as occurrence of the arrhythmia within the first 5 days after cardiac surgery. AF was considered to be present when an irregular rhythm was detected in the absence of P waves and/or presence an f wave
Perioperative myocardial infarction | In-hospital time, an average of 2 weeks
  Perioperative myocardial infarction was defined as an elevation in cardiac troponin accompanied by evidence of ischemia from ECG, angiographic, or imaging findings.
cardiac systolic function | within 5 days after surgery
  Improvement in either left ventricular ejection fraction or left ventricular end-systolic volume, as measured by echocardiography.
cardiac diastolic function | within 5 days after surgery
  Improvement in either E/e' ratio or left ventricular end-diastolic volume, as measured by echocardiography.
Abnormal blood potassium concentration | within 5 days after surgery
  blood potassium concentration<3.5mmol/L or >5.5mmol/L
postoperative blood glucose level | within 5 days after surgery
Inflammatory biomarkers | within 5 days after surgery
  high-sensitivity C-reactive protein, interleukin-1β, interleukin-6, interleukin-8, and tumor necrosis factor-α
Hs-Troponin-I | within 5 days after surgery
ICU stay | an average of 3 days
  ICU Stay was defined as the duration (in days) of initial postoperative stay in the intensive care unit following cardiac surgery.
Length of in-hospital time | an average of 2 weeks
  Length of in-hospital time was defined as the total number of days from the date of surgery to the date of hospital discharge.

OTHER OUTCOMES:
Safety Outcome | In-hospital time, an average of 2 weeks
  Diabetic ketoacidosis, severe hypoglycemic events, hypovolemia, urogenital tract infection, Incision infection and serious adverse events
ICU readmission | In-hospital time, an average of 2 weeks
  ICU readmission was defined as any unplanned readmission to the intensive care unit during the index hospitalization after the initial ICU discharge, regardless of cause.
Major adverse cardiac cerebrovascular events and its individual components | 30 days
  Major adverse cardiac cerebrovascular events composite includes all-cause mortality, myocardial infarction, stroke, and reoperation

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Zheng, MD,PhD, Principal Investigator — Fuwai Hospital, Chinese Academy of Medical Science
Locations (1):
- National Clinical Research Center for Cardiovascular Diseases, State Key Laboratory of Cardiovascular Disease, Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China